CLINICAL TRIAL: NCT05816018
Title: Improving Health Care in Major Depressive Disorder: a New Prognostic Tool Based on Gene Environment and Neuroimaging Signatures
Brief Title: Improving Health Care in Major Depressive Disorder
Acronym: DepType
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale San Raffaele (Other)
Collaborators: Ministry of Health, Italy (Other Government); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Benedetta Vai, Principal Investigator, Ospedale San Raffaele
Other Study IDs: GR-2019-12370616
Record Dates: First submitted 2023-03-14; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project aims to improve the health care provided to people with major depressive disorder (MDD), a disease which is a top cause of disability worldwide. One of the main obstacles to a more effective health care in these patients is represented by clinical heterogeneity, which has not completely elucidated biological correlates. Using a large sample of people with MDD already recruited (n=29,400), the investigators develop a clustering algorithm based on genetic-environmental and brain imaging predictors aimed at identifying homogeneous MDD subgroups. The researchers will then link these subgroups with relevant health outcomes, such as disease recurrency and severity, well-being and functioning, risk of psychiatric and medical comorbidities (e.g. cardiovascular disorders). Replication in independent samples already recruited(n=1380) will prove the validity of the subgroups and expand their clinical characterization. The investigators will develop a classification tool to link the individual's characteristics to the relevant health outcomes and provide corresponding clinical recommendations. The prognostic support tool will be applied to newly recruited samples, feasibility and usefulness according to clinicians's opinion will be assessed (n=120, ongoing recruitment).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of depressive episode in Major Depressive Disorder (DSM-5);
* at least one depressive episode preceding the current one;
* aged between 18 and 65;
* score of at least 8 on the Hamilton Depression Rating Scale (HDRS);
* signature of the information form and declaration of informed consent;
* elementary school certificate (as a minimum requirement for understanding the questions presented in the tests);
* native Italian speaker (or bilingualism).

Exclusion Criteria:

* diagnosis of bipolar disorder, cyclothymic disorder, schizophrenia and other psychotic spectrum disorders, neurodevelopmental disorders;
* diagnosis of intellectual disability, epilepsy, neurodegenerative disorders;
* disorders related to the use of drugs or alcohol in the last 6 months (except nicotine and caffeine);
* pregnant or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients and outpatients with an ongoing depressive episodes diagnosed accordingly to DSM 5.
Sampling Method: Non-Probability Sample
Enrollment: 30900 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
The depressive status | Assessment at the time of recruitment
  Assessment of the severity of disease using the Self-report Inventory Of Depressive Symptoms (IDS-SR) (Rush et al., 1996) with minimum-maximum values 0-116, higher scores mean a worse outcome, regarding the last week.
The self-report depressive symptomatology | Assessment at the time of recruitment
  Assessment of the depressive characteristics, using the Beck Depression Inventory (BDI) (Beck et al., 1961) with minimum-maximum values 0-39, higher scores mean a worse outcome, regarding the last 2 weeks.
The clinical evaluation of depressive symptomatology | Assessment at the time of recruitment
  Assessment of the presence of depressive status, Hamilton Depression Rating Scale (HDRS) (Hamilton, 1967) with minimum-maximum values 0-69, higher scores mean a worse outcome, regarding the current state.
The rate of cardiovascular and/or cardiometabolic diseases | Assessment at the time of recruitment
  Assessment of the presence/absence of lifetime and current cardiometabolic and/or cardiovascular diseases (e.g. diabetes, arterial hypertension, pulmonary arterial hypertension) based on extracted data from medical records and chart.

SECONDARY OUTCOMES:
The quality of functioning and well-being | Assessment at the time of recruitment
  Assessment of current and lifetime quality of life and well-being using the WHO Quality of Life-BREF (WHOQOL-BREF) (World Health Organization, 1996): the minimum and maximum values are 0-118, higher scores mean a better outcome, regarding the last 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Benedetta Vai, PhD, Principal Investigator — IRCCS San Raffaele Scientific Insititute
Locations (1):
- Benedetta Vai, Milan, Italy